CLINICAL TRIAL: NCT07395024
Title: A Phase 1 Crossover Design Study to Assess the Effect of CYP3A Moderate and Strong Inhibitors (Fluconazole and Itraconazole) and Strong Inducer (Carbamazepine) on the Single-dose Pharmacokinetics of ASP3082 in Healthy Adults
Brief Title: A Study to Learn How Fluconazole, Carbamazepine and Itraconazole Affect How the Body Processes ASP3082 in Healthy Adults
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 3082-CL-0102
Record Dates: First submitted 2026-01-28; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteer
Keywords: ASP3082; Pharmacokinetics; Setidegrasib; Healthy Volunteers; Fluconazole; Itraconazole; Carbamazepine
MeSH Terms: interventions — Fluconazole; Carbamazepine; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: ASP3082 + Fluconazole (Experimental): Participants receive ASP3082 on Days 1 and 15 and fluconazole on Days 8 to 28.
  Interventions: Drug: Setidegrasib; Drug: Fluconazole
- Group 2: ASP3082 + Carbamazepine (Experimental): Participants receive ASP3082 on Days 1 and 22 and carbamazepine on Days 8 to 28.
  Interventions: Drug: Setidegrasib; Drug: Carbamazepine
- Group 3: ASP3082 + Itraconazole (Experimental): Participants receive ASP3082 on Days 1 and 15 and itraconazole on Days 8 to 28.
  Interventions: Drug: Setidegrasib; Drug: Itraconazole

INTERVENTIONS:
Drug: Setidegrasib — Intravenous (IV) infusion
  Other Names: ASP3082
Drug: Fluconazole — Oral
  Arms: Group 1: ASP3082 + Fluconazole
Drug: Carbamazepine — Oral
  Arms: Group 2: ASP3082 + Carbamazepine
Drug: Itraconazole — Oral
  Arms: Group 3: ASP3082 + Itraconazole

SUMMARY:
Genes give your body instructions on how to make proteins. Proteins are needed to keep the body working properly. Many types of cancer are caused by changes in certain genes, making them faulty. Some people with solid tumors have a faulty KRAS gene. One such change in the KRAS gene is called a G12D mutation. Researchers are looking for ways to stop the actions of abnormal proteins made from the KRAS G12D mutation.

ASP3082 is thought to replace some of the abnormal proteins made from the faulty KRAS gene. If other medicines are given at the same time as ASP3082, they may affect how the body processes ASP3082.

In this study, fluconazole, itraconazole and carbamazepine are given with ASP3082 in healthy adults. The main aims are to check if fluconazole, itraconazole and carbamazepine affect how the body processes ASP3082. These medicines may affect how the body processes ASP3082 when they are taken at the same time.

This study will have 3 groups of adults. One group will be given fluconazole and ASP3082, the second group will be given carbamazepine and ASP3082, and the third group will be given itraconazole and ASP3082. ASP3082 will be given to people slowly through a tube into the vein (infusion). Fluconazole and carbamazepine will be given as a tablet and itraconazole will be given as a liquid by mouth. People will be given study treatments for about 1 month. They will then return to the clinic about 1 week after they finish study treatment for a final safety check.

ELIGIBILITY:
Inclusion Criteria:

* Participant is healthy and has no clinically significant medical condition based on the physical examination, electrocardiograms (ECGs) and protocol-defined clinical laboratory tests at screening or on day -1.
* Female participant is not pregnant and is not a woman of childbearing potential (WOCBP)
* Female participant must not be breastfeeding or lactating starting at screening and throughout the investigational period and for 5 half-lives (approximately 28 days after final study intervention administration).
* Female participant must not donate ova starting at first administration of study intervention and throughout the investigational period and for 3 months after final study intervention administration.
* Male participant must agree to use contraception with female partner(s) of childbearing potential (including breastfeeding partner) throughout the treatment period and for 3 months after final study intervention administration.
* Male participant must agree to remain abstinent or use a condom with pregnant partner(s) for the duration of the pregnancy throughout the investigational period and for 3 months after final study intervention administration.
* Male participant must not donate sperm during the treatment period and for 3 months after final study intervention administration.
* Participant agrees not to participate in another interventional study while participating in the present study.
* Participant has a Body Mass Index (BMI) range of 18.0 to 32.0 kg/m^2, inclusive, and weighs at least 50 kg at screening.

Exclusion Criteria:

* Participant is positive for Human Leukocyte Antigen (HLA) -B15:02 or HLA-A31:01, for Group 2 only.
* Participant has been pregnant within 6 months prior to screening.
* Participant has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease.
* Participant has a history of malignancy within 2 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that is considered cured with minimal risk of recurrence).
* Participant has had major surgery (e.g., requiring general anesthesia) within 90 days before screening, or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study or within 5 half-lives (approximately 28 days) after the last dose of study drug administration or end-of-study visit (ESV), whichever is longer.
* Participant has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 28 days prior to day -1.
* Participant has a history of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) DSM-5 criteria within 2 years before screening.
* Participant has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease or a family history of long QT syndrome.
* Participant has used any prescribed or nonprescribed drugs (including vitamins, and natural and herbal remedies, e.g., St. John's wort) in the 28 days prior to day -1, except for occasional use of acetaminophen (up to 2 g/day), topical dermatological products (including corticosteroid products) and hormone replacement therapy (HRT).
* Participant has used any inducer of metabolism (e.g., barbiturates and rifampin) in the 28 days prior to day -1.
* Participant has received a coronavirus disease 2019 (COVID-19) vaccine within the 14 days prior to day -1 or will have a COVID-19 vaccine dose before the ESV.
* Participant has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Participant has any liver test result alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST) or total bilirubin (TBL )) ≥ 1.5 ×upper limit of normal (ULN ) on day -1.
* Participant has a creatinine level outside normal limits on day -1.
* Participant has any of the following conditions on day -1: a mean pulse < 45 or > 90 bpm, mean systolic blood pressure (SBP ) > 140 mmHg, or mean diastolic blood pressure (DBP) > 90 mmHg (measurements taken in triplicate after participant has been resting in the supine position for at least 5 minutes; pulse measured automatically). If the mean blood pressure exceeds the limits above, 1 additional triplicate measurement may be taken.
* Participant has a mean corrected QT interval using Fridericia's formula (QTcF ) of > 450 msec on day -1.
* Participant tests positive for alcohol at screening or on day -1.
* Participant tests positive for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine and opiates) at screening or on day -1.
* Participant tests positive for cannabinoids on day -1.
* Participant has a positive serology test for hepatitis A virus (HAV) antibodies immunoglobulin M (IgM), hepatitis B (HBc) antibodies, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies or antibodies to human immunodeficiency virus (HIV ) type 1 and/or type 2 at screening.
* Participant has a positive rapid COVID-19 antigen test on day -1.
* Participant has any condition that makes the participant unsuitable for study participation.
* Participant has a known or suspected hypersensitivity to ASP3082 or any components of the formulation used.
* Participant has a history of smoking > 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to day -1 or the participant tests positive for cotinine at screening or day -1.
* Participant has a history of consuming > 10 units of alcoholic beverages per week within 3 months prior to screening (Note: 1 unit = 12 ounces of beer, 5 ounces of wine, 1.5 ounces of spirits/hard liquor).
* Participant has used any drugs of abuse (e.g., amphetamines, barbiturates, benzodiazepines, cocaine and/or opiates) within 3 months prior to day -1.
* Participant has had significant blood loss, donated ≥ 1 unit (450 mL) of whole blood or donated plasma within 7 days prior to day -1 and/or received a transfusion of any blood or blood products within 60 days prior to day -1.
* Participant has had previous exposure to ASP3082.
* Participant is an employee of Astellas, the study-related contract research organizations (CROs) or the clinical unit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of ASP3082 in plasma: Maximum Concentration (Cmax) in ASP3082 | Up to 29 days
  Cmax will be recorded from the PK plasma samples collected.
PK of ASP3082 in plasma: area under the concentration-time curve from time zero to the time of the last measurable concentration (AUClast) in ASP3082 | Up to 29 days
  AUClast will be recorded from the PK plasma samples collected.
PK of ASP3082 in plasma: area under the concentration-time curve extrapolated to infinity (AUCinf) in ASP3082 | Up to 29 days
  AUCinf will be calculated from the PK plasma samples collected.
PK of ASP3082 in plasma: Cmax in ASP3082+ Fluconazole (FLZ) | Up to 29 days
  Cmax will be recorded from the PK plasma samples collected.
PK of ASP3082 in plasma: AUClast in ASP3082+FLZ | Up to 29 days
  AUClast will be recorded from the PK plasma samples collected.
PK of ASP3082 in plasma: AUCinf in ASP3082+FLZ | Up to 29 days
  AUCinf will be calculated from the PK plasma samples collected.
Ratio of Cmax of ASP3082 and ASP3082+FLZ | Up to 29 days
  Ratios of Cmax will be calculated from the PK plasma samples collected.
Ratio of AUClast of ASP3082 and ASP3082+FLZ | Up to 29 days
  Ratios of AUClast will be calculated from the PK plasma samples collected.
Ratio of AUCinf of ASP3082 and ASP3082+FLZ | Up to 29 days
  Ratios of AUCinf will be calculated from the PK plasma samples collected.
PK of ASP3082 in plasma: Cmax in ASP3082+ Itraconazole (ITZ) | Up to 29 days
  Cmax will be recorded from the PK plasma samples collected.
PK of ASP3082 in plasma: AUClast in ASP3082+ITZ | Up to 29 days
  AUClast will be recorded from the PK plasma samples collected.
PK of ASP3082 in plasma: AUCinf in ASP3082+ITZ | Up to 29 days
  AUCinf will be calculated from the PK plasma samples collected.
Ratio of Cmax of ASP3082 and ASP3082+ITZ | Up to 29 days
  Ratios of Cmax will be recorded from the PK plasma samples collected.
Ratio of AUClast for ASP3082 and ASP3082+ITZ | Up to 29 days
  Ratios of AUClast will be recorded from the PK plasma samples collected.
Ratio of AUCinf for ASP3082 and ASP3082+ITZ | Up to 29 days
  Ratios of AUCinf will be calculated from the PK plasma samples collected.
PK of ASP3082 in plasma: Cmax in ASP3082+ Carbamazepine (CAR) | Up to 29 days
  Cmax will be recorded from the PK plasma samples collected.
PK of ASP3082 in plasma: AUClast in ASP3082+CAR | Up to 29 days
  AUClast will be recorded from the PK plasma samples collected.
PK of ASP3082 in plasma: AUCinf in ASP3082+CAR | Up to 29 days
  AUCinf will be calculated from the PK plasma samples collected.
Ratio of Cmax of ASP3082 and ASP3082+CAR | Up to 29 days
  Ratios of Cmax will be calculated from the PK plasma samples collected.
Ratio of AUClast for ASP3082 and ASP3082+CAR | Up to 29 days
  Ratios of AUClast will be calculated from the PK plasma samples collected.
Ratio of AUCinf for ASP3082 and ASP3082+CAR | Up to 29 days
  Ratios of AUCinf will be calculated from the PK plasma samples collected.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 36 days
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. NOTE: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. This includes events related to the comparator, if applicable, and events related to the (study) procedures.
Number of Participants with laboratory value abnormalities and/or AEs | Up to 36 days
  Number of participants with potentially clinically significant laboratory values.
Number of Participants with vital sign abnormalities and/or AEs | Up to 36 days
  Number of participants with potentially clinically significant vital sign values.
Number of Participants with electrocardiogram (ECG) abnormalities and/or AEs | Up to 36 days
  Number of participants with potentially clinically significant ECG values.
PK of FLZ in plasma: trough concentration (Ctrough) | Up to 25 days
  Ctrough of FLZ will be recorded from the PK samples collected.
PK of CAR in plasma Ctrough | Up to 28 days
  Ctrough of CAR will be recorded from the PK samples collected.
PK of ITZ in plasma Ctrough | Up to 25 days
  Ctrough of ITZ will be recorded from the PK samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.